CLINICAL TRIAL: NCT05883969
Title: Early Family-Centered Intervention for Infants With High-Risk of Cerebral Palsy: Protocol for the Randomized Controlled GO-PLAY Trial
Brief Title: GO-PLAY - Early Family-Centered Intervention for Infants With High-Risk of Cerebral Palsy
Acronym: GO-PLAY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Aalborg University Hospital (Other); Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Christina Høi-Hansen, Professor, MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-22041835
Record Dates: First submitted 2023-03-31; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early intervention for infants (Active Comparator): Early family-centered, individualized, goal-directed, intensive, and carried out within the home environment in a cross sectorial setting fortnightly contact shifting between at home visits and virtual meetings for 6 months after an interim diagnosis of CP or high risk of CP
  Interventions: Behavioral: GO-PLAY
- Usual care (Other): Standard care consists rehabilitation offered by the local hospital/community or other private initiatives when diagnosed with CP or high risk of CP. The approach, frequency, and location (at home or rehabilitation centers) is varied
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: GO-PLAY — The intervention is family-centered, individualized, goal-directed, intensive, and carried out within the home environment. The GO-PLAY intervention will last for six months and consists of a home visit once a month and a virtual meeting by telephone or video once a month. The intervention will be family centered. Experienced physiotherapists and occupational therapists will be the primary therapists providing the intervention to ensure uniformity. The motor learning element of the intervention is based on the principles of motor learning and dynamic systems theory. Emphasis is on children's self-initiated actions, which are stimulated by meaningful and motivating activities and toys. The child's play preferences to elicit self-generated motor activity will be the underlying basis of the training. Minimal manual guidance is provided when needed and withdrawn when the child demonstrates self-generated ability to complete part of the task.
  Arms: Early intervention for infants
Behavioral: Usual care — Children will receive referral for rehabilitation in the municipality as usual. Standard care consists of the additional follow up assessments in CP-EDIT as well as rehabilitation offered by their local hospital/community or other private initiatives when diagnosed with CP or high risk of CP. The approach, frequency, and location (at home or rehabilitation centers) is varied according to the center's protocol and not possible to standardize.
  Arms: Usual care

SUMMARY:
Background. Early diagnosis of cerebral palsy (CP) is important to enable appropriate intervention at a time when neuroplasticity is at its highest. Early intervention with focus on family-centered, home-based, parent-involved, and supervised by specialist therapists show positive cognitive and motor outcomes. This study adhere to international guidelines for early diagnosis and intervention, and include community therapists to ensure regular follow-up during and after the intervention period.

The aim of the current study is to compare the effectiveness of an early intervention program added to standard care, relative to standard care alone, on the early motor development in children from both a newborn and infant detectable risk pathway in a Danish multi-site setting.

Methods. In a randomized, controlled trial the response to the GO-PLAY (Goal Oriented ParentaL supported home ActivitY) intervention program added to standard care is superior to standard care alone is evaluated. The investigators will include infants from the Cerebral Palsy - Early Diagnosis and Intervention Trial (CP-EDIT registered separately at ClinicalTrials) and collect data at baseline, after intervention and at follow up when the children are 2 years corrected age.

The hypotheses are that the GO-PLAY intervention is more effective than standard care when the children are re-evaluated at the end of 6 months of intervention and that the parents involved in the GO-PLAY intervention will exhibit less signs of stress and anxiety and perceive the services that they are receiving as family-centered to a greater extent than parents of children receiving standard care.

Discussion. Approximately half of all infants with high risk of CP display high risk indicators identifiable by early screening before 5 months of age described as the newborn detectable risk pathway. The other half of all infants with CP are detected by parents, caregivers or health care professionals when displaying delayed motor milestones (e.g. hand asymmetry or not sitting at 9 months) and described as infant detectable risk pathway. There is a need to investigate if early intervention is effective in all infants with high suspicion of CP, also the ones with unremarkable neonatal history. Further, a systematic early intervention has not been tested in infants at high risk of CP in Denmark, where public health services include physiotherapy free of charge for infants with CP.

DETAILED DESCRIPTION:
Signs of CP may be visible already at three months of age but the mean diagnostic age is 13 months in Denmark. An early diagnosis is important in order to start relevant intervention when neuroplasticity is highest.

The study group will be recruited from the CP-EDIT, where both the newborn- and infant-detectable risk pathway from 3-12 months corrected age are included. Neonates may have obvious risk factors in the neonatal period, but in the present study infants with clinical findings suggesting CP emerging in the first year of life are also included. An interim diagnosis based on recommended predictive tools for early diagnosis; cerebral MRI, the General Movement Assessment (if < 5 months) and the Hammersmith Infant Neurological Examination will be an inclusion criteria for this study. In addition the Hand Assessment for Infants will be included to assess early hand asymmetry.

An estimated sample size of 60 participants in total; approximately 30 per group is expected. The infants will be allocated to groups based on stratified permuted block randomization: Stratification will be used to achieve an explicit balance for age in months (<6 months compared with ≥ 6 months) at study enrollment and gross motor development (HINE global score > 40 ambulant and ≤ 40 non ambulant). Eligible participants will be randomly assigned in permuted blocks of 2 and 6, according to computer-generated random numbers, to either GO-PLAY or standard care. The investigators anticipate that allocation concealment will be successful in preventing selection bias since the statistician conceal the allocation sequence from those assigning participants to the intervention groups, until the moment of assignment is disclosed; from which point the individual is part of the intention-to-treat (ITT) population.

The infants will be assessed on the occasions; at baseline, post intervention and follow up at 24 months corrected age

ELIGIBILITY:
Inclusion Criteria:

Infants will be included in the intervention study, if they fulfil at least one of the requirements A or B:

A. any two of the following:

* Neuroimaging predictive of a motor disability including the involvement of one or more of the following structures: sensori-motor cortex, basal ganglia, posterior limb of the internal capsule, pyramidal tracts.
* General Movement Assessment with absent fidgety GMs at fidgety age
* HINE scores <57 at 3months or <60 at 6months or <63 at 9 months or <66 at 12 months

B. both of the following:

* Unilateral brain injury on neuroimaging (MRI or ultrasound) predictive of CP
* Clinical signs of asymmetry

Exclusion Criteria:

* Infants with progressive or neurodegenerative disorders or genetic disorders not associated with CP
* Infants with other disability diagnoses e.g. Down Syndrome.
* children for whom neither parent is fluent in Danish.

Ages: 3 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Peabody Developmental Motor Scales - Second edition (PDMS-2) | Change from baseline at 6 months
  PDMS-2 is a standardized, norm-referenced measure used to evaluate the gross and fine motor development of children aged birth to 6 years. The gross motor component is comprised of four subtests: reflexes (raw score range 0-16), stationary (raw score range 0-60), locomotion (raw score range 0-178) and object manipulation (raw score range 0-48). Two subtests, grasping (raw score range 0-52) and visual-motor integration (raw score range 0-144), form the fine motor component. The total Motor Quotient (TMQ) is formed by a combination of the results of the gross and fine motor subtests. The PDMS-2 TMQ range from 90-165 (indicating average or above average age-normed motor abilities) to 89-35 (indicating below average to very poor age-normed motor abilities).

SECONDARY OUTCOMES:
Alberta Infant Motor Scale (AIMS) | Change from baseline at 6 months
  AIMS is an observational assessment scale constructed to measure gross motor maturation in infants from birth through independent walking. 58 items are generated and organized into four positions: prone, supine, sitting and standing. Each item describes three aspects of motor performance weight-bearing, posture and antigravity movements. The overall score ranges from a minimum of 0 to a maximum of 58.
Gross Motor Function Measure (GMFM-66) | Change from baseline at 6 months (if > 5 months at inclusion)
  GMFM-66 is a criterion-referenced tool designed and evaluated to measure changes in gross motor function over time or with intervention in children with CP. It consists of 5 dimensions rolling, sitting, walking, running, and jumping. The 66 items are organized in increasing difficulty order from 0 (low capacity) to 100 (high capacity) along an interval scale. Each item is scored on a four-point Likert scale (0-3). It can be used from 5 months of age, and a 5- year-old typically developing child is expected to achieve a score of 100.
Hand Assessment in Infants (HAI) | Change from baseline at 6 months (if<12 months)
  HAI is an assessment developed for infants at risk of developing CP in the age range 3-12 months. The test procedure comprises a semi-structured video-recorded play session lasting 10- 15 min. A test kit of toys is presented to the infant to encourage and elicit exploration, making a wide range of a unilateral and bilateral hand movements observable. The HAI measures the degree and quality of goal directed actions performed with each hand separately as well as both hands together. It provides a separate score for each hand (Each Hand Sum Score 0-24), a score for both hands (Both Hands Sum Score 0-58), an asymmetry index in % illustrating possible asymmetric hand use as well as criterion referenced measure of general upper limb ability (HAI-units 0-100)
The Parental Stress scale (PSS) | Change from baseline at 6 months
  PSS is an 18-item questionnaire assessing parents' feelings about their parenting role, exploring both positive (emotional benefits, personal development) and negative aspects (demands on resources, feelings of stress) of parenthood. The overall score ranges from a minimum of 18 to a maximum of 90
The Depression Anxiety Stress Scales (DASS-21) | Change from baseline at 6 months
  DASS-21 is an adult self-report designed to measure the emotional states of depression, anxiety and stress. It is a 4221-item questionnaire and will be used to measure parent emotional well-being
The Measure of Processes of Care 20 (MPOC-20) | 6 months post baseline
  MPOC-20 is a self-report measure of parents' perceptions of the extent to which the health services they and their child(ren) receive are family-centered. The 20 items consist of 5 domains; enabling and partnership, providing general information, providing specific information about the child, respectful and supportive service, and coordinated and comprehensive care.

OTHER OUTCOMES:
Peabody Developmental Motor Scales - Second edition (PDMS-2) | at 24 months corrected age
  PDMS-2 is a standardized, norm-referenced measure used to evaluate the gross and fine motor development of children aged birth to 6 years. The gross motor component is comprised of four subtests: reflexes (raw score range 0-16), stationary (raw score range 0-60), locomotion (raw score range 0-178) and object manipulation (raw score range 0-48). Two subtests, grasping (raw score range 0-52) and visual-motor integration (raw score range 0-144), form the fine motor component. The total Motor Quotient (TMQ) is formed by a combination of the results of the gross and fine motor subtests. The PDMS-2 TMQ range from 90-165 (indicating average or above average age-normed motor abilities) to 89-35 (indicating below average to very poor age-normed motor abilities).
Gross Motor Function Measure (GMFM-66) | at 24 months corrected age
  GMFM-66 is a criterion-referenced tool designed and evaluated to measure changes in gross motor function over time or with intervention in children with CP. It consists of 5 dimensions rolling, sitting, walking, running, and jumping. The 66 items are organized in increasing difficulty order from 0 (low capacity) to 100 (high capacity) along an interval scale. Each item is scored on a four-point Likert scale (0-3). It can be used from 5 months of age, and a 5- year-old typically developing child is expected to achieve a score of 100.
Bayley Scales of Infant and Toddler Development 4 (BSID-4) -cognitive | at 24 months corrected age
  BSID-4 is a standardized and norm-referenced assessment, which measures the cognitive, motor, language and social-emotional development of infants and toddlers aged 0-3. Raw scores of successfully completed items are converted to scale scores and to composite scores. These scores are used to determine the child's performance compared with norms taken from typically developing children of the same age.
The Ages & Stages Questionnaire (ASQ-3) | at 24 months corrected age
  ASQ-3 pinpoints developmental progress in children between the age of one month to 5 ½ years. It has a parent-centric approach and is used as a developmental screener
The Parental stress scale (PSS) | at 24 months corrected age
  PSS is an 18-item questionnaire assessing parents' feelings about their parenting role, exploring both positive (emotional benefits, personal development) and negative aspects (demands on resources, feelings of stress) of parenthood. The overall score ranges from a minimum of 18 to a maximum of 90
The Depression Anxiety Stress Scales (DASS-21) | at 24 months corrected age
  DASS-21 is an adult self-report designed to measure the emotional states of depression, anxiety and stress. It is a 21-item questionnaire and will be used to measure parent emotional well-being
The Measure of Processes of Care 20 (MPOC-20) | at 24 months corrected age
  MPOC-20 is a self-report measure of parents' perceptions of the extent to which the health services they and their child(ren) receive are family-centered. The 20 items consist of 5 domains; enabling and partnership, providing general information, providing specific information about the child, respectful and supportive service, and coordinated and comprehensive care.
Measure of Processes of Care-Service Provider (MPOC-SP) | 6 months post baseline
  MPOC-SP are used to measure the experiences of health care providers working with children with long-term health or developmental difficulties, and their families. The MPOC-SP has 27-items covering four scales. All response options are labelled, ranging from 1 ("never") to 7 ("to a great extent"). A higher score indicates that the service provider evaluates the service as family-centred.
Measure of Processes of Care-Service Provider (MPOC-SP) | at 24 months corrected age
  MPOC-SP are used to measure the experiences of health care providers working with children with long-term health or developmental difficulties, and their families. The MPOC-SP has 27-items covering four scales. All response options are labelled, ranging from 1 ("never") to 7 ("to a great extent"). A higher score indicates that the service provider evaluates the service as family-centred.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Hoi-Hansen, Professor, Study Chair — Department of Paediatrics, University Hospital Rigshospitalet, Denmark
Locations (2):
- Denmark (2):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus